CLINICAL TRIAL: NCT04093193
Title: The Efficacy of Debridement of the Sinus Cavity Following Primary Functional Endoscopic Sinus Surgery (FESS): A Randomized Controlled Trial.
Brief Title: Debridement and Functional Endoscopic Sinus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Director, St. Paul's Sinus Centre, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H15-02071
Record Dates: First submitted 2019-06-07; First posted 2019-09-17 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: Functional Endoscopic Sinus Surgery
MeSH Terms: conditions — Disease | interventions — Debridement

STUDY DESIGN:
Intervention Model Description: There will be two possible scenarios resulting from randomization:
  1. The patient is randomized to the arm that receives routine post-operative debridement (treatment group).
  2. The patient is randomized to the arm that will not receive post-operative debridement (control group).
Who Masked: Investigator
Masking Description: The patient will know if he/she is getting debridement or not. The PI will comment on all the objective outcome measures and will be the blinded assessor (he will not perform the debridements).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Debridement group (Experimental): Patients receive routine post-operative debridement at their Day 6, 30 and 60 follow up appointments.
  Interventions: Procedure: Debridement
- Non Debridement Group (No Intervention): Patients will not receive debridement at any follow up visit after surgery. They will continue with saline irrigation.

INTERVENTIONS:
Procedure: Debridement — Debridement or cleaning of the sinuses post-operatively has been described as a regular post-surgery procedure .
  Arms: Debridement group

SUMMARY:
Functional endoscopic sinus surgery (FESS) is the gold standard surgical intervention for management of patients with chronic rhinosinusitis (CRS). Synechiae formation in the middle meatus is the most common complication of endoscopic sinus surgery after FESS. Nasal debridement is a postoperative procedure used in the prevention of synechiae formation. This procedure lacks standardized evidence-based guidelines. The currently existing studies that have been conducted to determine the efficacy of post-operative debridement have shown conflicting results. We hypothesize that there is no difference in short and long term clinical outcomes between patients who had routine post-operative nasal debridement following FESS and patients who did not have post-operative nasal debridement.

DETAILED DESCRIPTION:
Purpose The purpose of this study is to assess the efficacy of post-FESS nasal debridements in the prevention of post-operative synechiae formation.

Hypothesis There is no difference in short and long term clinical outcomes between patients who had routine post-operative nasal debridement following FESS and patients who did not have post-operative nasal debridement.

Justification To prevent synechiae formation, many studies have been published evaluating the efficacy of post-operative debridement procedures. Many of these studies have shown conflicting results. There were many inconsistent variables between the studies, such as limited follow-up periods, varying extent of surgery, and variability in pre and post-operative treatment.

With a well designed study, we would like to assess if there is a difference in the incidence of formation of middle meatal synechiae between patients who have debridement and patients who don't.

This will further add much needed evidence to the need for this procedure in the post operative period following FESS.

Surgery The participants in this study will all undergo standard-of-care functional endoscopic sinus surgery (FESS) to treat their sinus disease. No changes will be made to pre-operative or operative protocol on account of this study. All post-operative standard-of-care procedures and medication will be maintained.

Follow up visits After FESS, participant subjects will be asked to return for 4 follow-up visits within the first 90 days and one follow-up visit at 180 days. They will be asked to return at 6, 30, 60, 90 and 180 days following their sinus surgery. At their 6 and 30 day follow-up visits they will either receive or not receive routine post-operative debridement depending on randomization.

Statistical Analysis

Sample size calculations A sample size calculation was performed to determine the appropriate number of patients required to adequately compare the incidence of synechiae between participants with versus without postoperative debridement following FESS. Previous investigations at the St. Paul's Sinus Centre have found that of post-FESS cases, 18% develop synechiae from use of gloved-Merocel middle meatal spacers. Utilizing a type I error of 5%, type II error of 20%, effect difference of 15% and 10% loss to follow-up, a total of 150 patients are required (75 per arm).

Statistical Comparisons The primary objective of this randomized controlled trial will be to compare the incidence of synechiae between subjects receiving debridement versus those receiving saline irrigation (no debridement) up to 180 days post-surgery. Count and absolute percentages of synechia incidence will be reported. The Chi-Squared test will be used to determine statistical significance between incidence rates. Probability values less than 5% (α=0.05) will be considered significant. Corresponding odds ratios and 95% confidence intervals will be reported.

For the secondary outcome measures (e.g. Sinonasal Outcomes Test 22 SNOT-22, PJESS/MLK), results will be summated and considered as continuous, numerical variables. Descriptive statistics using mean, median, standard deviation and inter-quartile ranges will be reported. The unpaired two sample student t-tests will be applied to investigate the difference between the means of the various outcome measures. Probability values less than 5% (α =0.05) will also be considered statistically significant.

Baseline demographics and clinical factors will be compared between each treatment group to determine whether randomization yielded comparable groups. Multivariable logistic and linear regression will be used to investigate the relationship between postoperative debridement and the primary (incidence of synechiae) or secondary outcomes (PJESS/MLK).

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 19;
* Have chronic sinus disease (CRS) and are scheduled to undergo sinus surgery on both sides of your nose for the first time.

Exclusion Criteria:

* Unable to speak English;
* Are having surgery for the removal of a nasal tumor;
* Have a disorder of your immune system in which your body's immune system attacks itself (autoimmune disorder)
* Diagnosed with cystic fibrosis
* Have had sinus surgery in the past
* Are scheduled to have a procedure known as nasal septal reconstruction, without additional sinus surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-06-22 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Postoperative Synechiae | Day 30, 60, 90, and 180 follow-up visits.
  The existence of postoperative synechiae will be considered as a categorical, dichotomous outcome variable (presence or absence).

SECONDARY OUTCOMES:
Sinonasal Outcomes Test - 22 (SNOT-22) | Day 30, 60, 90, and 180 follow-up visits.
  The SNOT-22 is a sinus-specific questionnaire that evaluates subjective symptoms for patients suffering from chronic rhinosinusitis.
  SNOT-22 is scored out of 110 (22 questions, up to 5-points each) has demonstrated internal consistency, reliability, discriminate and concurrent validity and responsiveness to change. Responses will be summated and considered as a continuous, numerical variable.
Philpott-Javer (PJ) and Modified Lund-Kennedy (MLK) Endoscopic Staging System (ESS) | Day 30, 60, 90, and 180 follow-up visits.
  Sinonasal mucosal inflammation is an objective measure assessed endoscopically and graded on both the PJ and MLK ESS for CRS.
Visual Analog Score (VAS) for pain and discomfort | Day 6, 30, 60, 90, and 180 follow-up visits.
  The visual analog score describes subjective pain and discomfort levels experienced by the participant following the procedures in both arms of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- E.N.T Clinic, St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available to other researchers.

REFERENCES:
- [Background] Bachert C, Pawankar R, Zhang L, Bunnag C, Fokkens WJ, Hamilos DL, Jirapongsananuruk O, Kern R, Meltzer EO, Mullol J, Naclerio R, Pilan R, Rhee CS, Suzaki H, Voegels R, Blaiss M. ICON: chronic rhinosinusitis. World Allergy Organ J. 2014 Oct 27;7(1):25. doi: 10.1186/1939-4551-7-25. eCollection 2014. PMID 25379119
- [Background] Fernandes SV. Postoperative care in functional endoscopic sinus surgery? Laryngoscope. 1999 Jun;109(6):945-8. doi: 10.1097/00005537-199906000-00020. PMID 10369288
- [Background] Green R, Banigo A, Hathorn I. Postoperative nasal debridement following functional endoscopic sinus surgery, a systematic review of the literature. Clin Otolaryngol. 2015 Feb;40(1):2-8. doi: 10.1111/coa.12330. PMID 25314101
- [Background] Bednarski KA, Kuhn FA. Stents and drug-eluting stents. Otolaryngol Clin North Am. 2009 Oct;42(5):857-66, x. doi: 10.1016/j.otc.2009.07.001. PMID 19909864
- [Background] Miller RS, Steward DL, Tami TA, Sillars MJ, Seiden AM, Shete M, Paskowski C, Welge J. The clinical effects of hyaluronic acid ester nasal dressing (Merogel) on intranasal wound healing after functional endoscopic sinus surgery. Otolaryngol Head Neck Surg. 2003 Jun;128(6):862-9. doi: 10.1016/S0194-59980300460-1. PMID 12825038
- [Background] Saafan ME, Ragab SM, Albirmawy OA, Elsherif HS. Powered versus conventional endoscopic sinus surgery instruments in management of sinonasal polyposis. Eur Arch Otorhinolaryngol. 2013 Jan;270(1):149-55. doi: 10.1007/s00405-012-1969-8. Epub 2012 Apr 10. PMID 22487908
- [Background] Catalano PJ, Roffman EJ. Evaluation of middle meatal stenting after minimally invasive sinus techniques (MIST). Otolaryngol Head Neck Surg. 2003 Jun;128(6):875-81. doi: 10.1016/S0194-59980300469-8. PMID 12825040
- [Background] Jorissen M. Postoperative care following endoscopic sinus surgery. Rhinology. 2004 Sep;42(3):114-20. PMID 15521662
- [Background] Lund VJ, MacKay IS. Outcome assessment of endoscopic sinus surgery. J R Soc Med. 1994 Feb;87(2):70-2. doi: 10.1177/014107689408700204. No abstract available. PMID 8196032
- [Background] Stammberger H. Endoscopic endonasal surgery--concepts in treatment of recurring rhinosinusitis. Part I. Anatomic and pathophysiologic considerations. Otolaryngol Head Neck Surg. 1986 Feb;94(2):143-7. doi: 10.1177/019459988609400202. PMID 3083326
- [Background] Kennedy DW. Prognostic factors, outcomes and staging in ethmoid sinus surgery. Laryngoscope. 1992 Dec;102(12 Pt 2 Suppl 57):1-18. PMID 1453856
- [Background] Bugten V, Nordgard S, Steinsvag S. The effects of debridement after endoscopic sinus surgery. Laryngoscope. 2006 Nov;116(11):2037-43. doi: 10.1097/01.mlg.0000241362.06072.83. PMID 17075402
- [Background] Bugten V, Nordgard S, Steinsvag S. Long-term effects of postoperative measures after sinus surgery. Eur Arch Otorhinolaryngol. 2008 May;265(5):531-7. doi: 10.1007/s00405-007-0501-z. Epub 2007 Oct 25. PMID 17960410
- [Background] Alsaffar H, Sowerby L, Rotenberg BW. Postoperative nasal debridement after endoscopic sinus surgery: a randomized controlled trial. Ann Otol Rhinol Laryngol. 2013 Oct;122(10):642-7. PMID 24294687
- [Background] Nilssen EL, Wardrop P, El-Hakim H, White PS, Gardiner Q, Ogston S. A randomized control trial of post-operative care following endoscopic sinus surgery: debridement versus no debridement. J Laryngol Otol. 2002 Feb;116(2):108-11. doi: 10.1258/0022215021910041. PMID 11827582
- [Background] Lee JY, Byun JY. Relationship between the frequency of postoperative debridement and patient discomfort, healing period, surgical outcomes, and compliance after endoscopic sinus surgery. Laryngoscope. 2008 Oct;118(10):1868-72. doi: 10.1097/MLG.0b013e31817f93d3. PMID 18641526